CLINICAL TRIAL: NCT03697291
Title: Comparison of the Self-invented Intracavitary ECG Wire With the Commercial System - Certodyn®
Brief Title: Self-invented Intracavitary ECG Wire VS the Commercial System - Certodyn®
Acronym: iECG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Prasert Sawasdiwipachai, Principal investigator, Mahidol University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Si 548/2018
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Central Line Complication
Keywords: Self invented iECG wire; PS wire; Certodyn; intracavitary ECG; PICC line; giant P wave

STUDY DESIGN:
Intervention Model Description: Single center, prospective, cross over study
Who Masked: Outcomes Assessor
Masking Description: unlabeled ECG print
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS wire (Experimental): self-invented iECG wire
  Interventions: Device: PS wire
- Certodyn (Active Comparator): Commercially available iECG system - Certodyn
  Interventions: Device: PS wire

INTERVENTIONS:
Device: PS wire — The wiring connection used to convey ECG signal from inside the body
  Other Names: Self-invented iECG wire

SUMMARY:
Peripherally Inserted Central Catheter (PICC) is considered a central venous line placement (CVL) which mandates the confirmation of the tip's location. At present, most CVL's position are confirmed by radiographic method either by in-procedure fluoroscopy or post-insertion x-ray. For CVLs placed from upper body (from internal jugular vein, subclavian veins or upper arm veins), the intracavitary electrocardiogram (iECG) can also be used.

Intracavitary ECG are proven effective for tip confirmation and provide some benefits i.e. lower cost, decrease exposure to harmful radiation for care providers and also the patients, require less personals and equipments, provide real-time confirmation as comparable to fluoroscopy, etc. There are several devices and makes of iECG apparatus but B.Braun-Certodyn® remains the only available system in our institution. The limitation is the availability of the Certodyn devices on each locations where CVL will be placed i.e. operating theater, intensive care unit, bedside placement, radiology suite, etc. Since the connecting wire is only supplied in the certain CVL kits under B.Braun brand, this has rendered iECG for other types or makes of CVL or PICC line become even more difficult.

Self-invented connector wire for iECG (PS wire) has been made and used effectively in the past few years at Siriraj hospital. The patent registration is underway and the author seek to compare this PS wire against the commercial Certodyn system.

DETAILED DESCRIPTION:
Objective

1. To evaluate the success rate of iECG CVL tip confirmation by self-invented iECG connector wire.
2. To compare quality of iECG tracing produced from both of self-invented iECG wire versus the Certodyn system.

Materials, participants and study method

Equipments required:

1) Self-invented iECG wire (PS wire) 2) Commercial iECG system which consists of the Certodyn and the wire. 3) Standard ECG monitoring system which can display and printout the ECG tracing. 4) A digital ECG caliper which can measure P wave amplitude and noise segment in millimeter up to 2 decimal points. Study method

1. Patient presented for PICC line from upper torso will be screened and assessed for eligibility.
2. Exclusion criteria includes children younger than 18 yo, patient with atrial fibrillation or other rhythms not generated from intrinsic SA node i.e. pacer, unstable hemodynamic, patient with history arrhythmias, HR > 120 bpm, patients with hypercoagulable state, allergy to heparin or patients with known heparin induced thrombocytopenia, patients with known Creutzfeldt-Jakob Disease
3. Obtain informed consent.
4. Patient will be monitored with standard 3-lead ECG, the baseline lead II ECG will be printed out and tagged with a serial number.
5. Patient will undergo the standard PICC line placement using Seldinger or modified Seldinger technique. The catheter will be pre-flushed with 10 units/mL heparinized NSS. When catheter is inserted into the proximal SVC (guided by landmark measurement), the wire will be retracted to the marked location where the tip of the wire is at the end of the catheter. The iECG connection by Certodyn will be applied. The catheter and wire will be adjusted until the giant P wave (highest P) was detected on screen, this ECG tracing will be printed out and tagged with another non-sequential serial number. The iECG will then switched to the PS wire and the iECG tracing will be printed out again and tagged with another non-sequential serial number. All 3 ECG printouts will be stapled together for measurement by cardiologist who is blind to the intervention later.
6. The intervention related to research study is considered ended at this point. The patient will have their CVL/PICC line adjusted to the proper position (mid to distal SVC for mid-long term and long term catheter). The CVL or PICC will be secured, flushed and locked per standard protocol.
7. Portable CXR will be routinely obtained when patients arrived to the ward. The information of the tip of the catheter will be recorded as well.

Data analysis

1. Demographic data, type of catheter, depth of catheter where giant P wave obtained and final position of catheter will be recorded.
2. Each study patient produce 3 ECG print outs which are -baseline surface lead II ECG

   * iECG produced by Certodyn system
   * iECG produced by PS wire Each ECG tracing will be evaluated and measured by a cardiologist who is blind to the intervention. The 2 measured parameters includes:
   * The amplitude of P wave in mm from baseline surface ECG of each cardiac cycle. -The amplitude of giant P wave in mm from iECG from both Certodyn and PS wire.
3. All 3 ECG print outs will be compared for quality and the length noisy ECG segment (determined as the ECG with interference artifact of baseline > 1 mm) will also be measured in mm.

6) All measurement will be analyzed statistically to determine the differences between the 2 systems.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years and above.
* Requires PICC line insertion from upper torso.

Exclusion Criteria:

* Children younger than 18 years.
* Patient with atrial fibrillation or other rhythms not generated from intrinsic SA node i.e. pacer, atrial fibrillation, etc.
* Unstable hemodynamic.
* Patient with history arrhythmias.
* Patient with HR > 120 bpm.
* Patients with hypercoagulable state.
* Allergy to heparin.
* Patients with known heparin induced thrombocytopenia.
* Patients with known Creutzfeldt-Jakob Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Signal noise ratio | 10 minutes
  Measuring the segment of ECG noise (if exists) in millimeters compare to the total ECG segment. Compare this signal noise ratio between the baseline surface ECG, the self-invented wire derived iECG and the Certodyn derived iECG.

SECONDARY OUTCOMES:
The amplitude of giant P Wave | 5 minutes
  Measure the amplitude of each giant P wave obtained from ECG print out from iECG derived from both certodyn and self-invented iECG wire.

CONTACTS AND LOCATIONS:
Overall Officials: Prasert Sawasdiwipachai, MD, Principal Investigator — Anesthesiology department Siriraj hospital
Locations (2):
- Thailand (2):
  - Siriraj hospital, Mahidol university, Bangkok Noi, Bangkok
  - Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Oster, D.D. "Improving ECG trace quality." Biomedical Instrumentation & Technology, 2000; 34: 219-222. 2. Corsten SA, van Dijk B, Bakker NC, de Lange JJ, Scheffer GJ. Central venous catheter placement using the ECG-guided Cavafix-Certodyn SD catheter. J Clin Anesth. 1994; 6(6): 469-72. 3. Pittiruti M, La Greca A, Scoppettuolo G. The electrocardiographic method for positioning the tip of central venous catheters. J Vasc Access. 2011; 12(4): 280-91. 4. Pittiruti M, Bertollo D, Briglia E, Buononato M, Capozzoli G, De Simone L, La Greca A, Pelagatti C, Sette P. The intracavitory ECG method for positioning the tip of central venous catheters: results of an italian multicenter study. J Vasc Access. 2012; 13(3):357-65. 5. Wang G, Guo L, Jiang B, Huang M, Zhang J, Qin Y. Factors Influencing Intracavitory Electrocardiographic P-Wave Changes during Central Venous Catheter Placement. PLoS One. 201510(4):e0124846. 6. Yuan L, Li R, Meng A, Feng Y, Wu X, Yang Y, et al. Superior success rate of intracavitory electrocardiogram guidance for peripherally inserted central catheter placement in patients with cancer: A randomized open-label controlled multi center study. PLoO One. 2017; 12(3):e0171630.